CLINICAL TRIAL: NCT06916559
Title: Novel Derivatization-Based HPLC for Urinary Oxalate and Citrate: A Superior Clinical Alternative to Ion Chromatography
Brief Title: Comparison of Different Methods for Measuring Urinary Oxalate and Citrate: An Observational Study
Acronym: Comparison of
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice-President, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: ES-2024-242-01
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hyperuricosuria; Hypocitraturia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Urolithiasis
- Healthy people

SUMMARY:
This observational study aims to compare three different laboratory methods for measuring urine oxalate and citrate concentrations. The primary objective is to evaluate whether an improved High-Performance Liquid Chromatography (HPLC) method-using a novel derivatization reagent-can achieve similar accuracy to the gold standard Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) while offering advantages in cost, speed, and ease of use in routine clinical settings.

The study will involve the collection of morning urine samples from both healthy volunteers and patients with urolithiasis (urinary stones). Each urine sample will be tested using the following three methods:

1. Modified High-Performance Liquid Chromatography (HPLC): This method builds on traditional HPLC technology by incorporating a novel derivatization reagent to enhance the sensitivity and accuracy of detecting oxalate and citrate. The improved HPLC method is designed to be less time-consuming and more cost-effective, which could make it a viable option for regular clinical use.
2. Ion Chromatography (IC): Widely used in many hospital laboratories, the IC method detects urine oxalate and citrate without the need for a derivatization step. While this method is straightforward and convenient, its sensitivity and accuracy are expected to be lower compared to LC-MS/MS and the modified HPLC method.
3. Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS): LC-MS/MS is currently considered the gold standard for measuring urine oxalate and citrate due to its high sensitivity and specificity. However, the method requires expensive equipment and involves complex procedures, limiting its routine application in most clinical laboratories.

Participants will provide urine samples, which will be divided and analyzed using all three methods simultaneously. The study will assess the correlation and consistency between the methods, with a particular focus on comparing the modified HPLC method to LC-MS/MS. Statistical analyses, including Bland-Altman analysis and linear regression, will be used to determine the agreement between the measurement techniques.

This study is non-interventional and involves only the collection of urine samples, posing minimal risk to participants. Informed consent will be obtained from all participants after they are fully briefed about the study objectives, procedures, and any potential risks. All collected data will be managed confidentially and analyzed rigorously to ensure the reliability of the findings.

If the modified HPLC method demonstrates comparable accuracy to LC-MS/MS, it could provide a more accessible, cost-effective, and timely option for routine clinical measurement of urinary oxalate and citrate. Such an improvement in laboratory diagnostics may support better clinical decision-making in the prevention and management of urinary stone disease, ultimately benefiting patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging evidence indicating the presence of urinary stones (stone patient group).
2. Imaging evidence indicating the absence of urinary stones (control group).

Exclusion Criteria:

1. Patients who are unable to understand or complete the study documentation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This observational study will enroll adult participants from two groups: patients with urolithiasis (specifically those exhibiting hyperuricosuria and hypocitraturia) and healthy volunteers without any history of urinary stone disease or related metabolic disorders. The study aims to compare urinary uric acid and citrate measurements obtained using three different analytical methods.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Uric Acid Measurements from Three Methods | Baseline sample analysis, with all measurements completed within 24 hours of sample collection.
  The primary outcome is to compare the uric acid measurement results obtained from three analytical methods: modified High-Performance Liquid Chromatography (HPLC) using a novel derivatization reagent, Ion Chromatography (IC), and Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS). This outcome will be evaluated by determining the mean differences, 95% confidence intervals, and correlations among the three methods using Bland-Altman analysis and linear regression. The goal is to assess whether the modified HPLC method can reliably reflect uric acid levels comparable to the LC-MS/MS gold standard.

SECONDARY OUTCOMES:
Comparison of Urinary Citrate Measurements from Three Methods | Baseline sample analysis, with all measurements completed within 24 hours of sample collection.
  The secondary outcome is to evaluate and compare the urinary citrate concentration results obtained from the three methods: modified HPLC, Ion Chromatography (IC), and LC-MS/MS. The analysis will include calculating mean differences, 95% confidence intervals, and assessing the degree of correlation among the methods using statistical tools such as Bland-Altman plots and linear regression. This outcome will help determine the consistency and reliability of citrate measurements across the different analytical techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Guangdong Key Laboratory of Urology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No